CLINICAL TRIAL: NCT07375810
Title: A Study to Measure Underlying Coronary Stenosis; a Prospective, Multi-Center Study to Measure Efficacy of ECGio Against Multiple Reference Standards
Brief Title: Analysis of ECGio to Predict Coronary Stenosis Against a Mixed Reference Standard
Acronym: SUPER
Status: Not yet recruiting | Type: Observational
Sponsor: Heart Input Output Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HIO0004A
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Artificial Intelligence; Electrocardiogram; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- CT Angiogram: This is the Cohort which received only Computed Tomography Angiography as a part of the study
- Invasive Angiography: This is the Cohort which received both Computed Tomography Angiography and Invasive Angiography as a part of the study
- Enrollment Period 2: This Cohort is the continuation of enrollment of invasive angiogram patients beyond the completion of the primary endpoint

SUMMARY:
The study objective is to evaluate the effectiveness of the ECGio algorithm in predicting clinically significant coronary artery disease . ECGio's diagnostic performance during the trial will be compared against an objective performance ¬criteria using a mixed reference standard of quantitative coronary angiography and quantitative coronary computed tomography angiography in patients a general adult population under suspicion of coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older at time of data collection.
2. Patients with medical records stored in a digitized format.
3. Patients under suspicion of coronary artery disease (both suspicion of significant coronary artery disease as well as to rule out significant CAD) who present to the site with an electrocardiogram recorded up to 30 days prior to Coronary Computed Tomography Angiography.

Exclusion Criteria:

1. Patients with acute coronary syndrome.
2. Patients who previously underwent coronary artery bypass grafting.
3. Patients whose electrocardiogram tracing has extreme noise or artifact to the extent that it would be recommended to redo the tracing.
4. Patients with prior percutaneous coronary intervention resulting in stenting.
5. Unanalyzable invasive coronary angiogram.
6. Unanalyzable Coronary Computed Tomography Angiography.
7. Unanalyzable electrocardiogram signal.
8. Incomplete invasive coronary angiogram (e.g., only the right coronary artery was injected and visualized).
9. Patient core lab analyzed Coronary Computed Tomography Angiography showed ≥ 50% blockage in any vessel but patient was not referred to invasive coronary angiogram.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be made up of all-comers to Coronary Computed Tomography Angiography from each site taking up to the first 250, consecutive patients recruited for the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 978 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity & Specificity | Within 30 days of enrollment
  The lower 95% bound of ECGio's sensitivity and specificity in patients who underwent invasive angiography or computed tomography angiography (Co-primary endpoints)

SECONDARY OUTCOMES:
Sensitivity & Specificity | For the first 300 patients referred to invasive angiography through study completion, an average of 90 days
  The lower 95% bound of ECGio's sensitivity and specificity in patients who underwent invasive angiography (Co-secondary endpoints) in enrollment period 2
Demographic Performance | For patients in the 30 days following computed tomography angiography
  ECGio's predictive performance across different demographic groups (e.g Race, Sex, Risk Factors)
Angiographic Stenosis Prediction | For the first 300 patients referred to invasive angiography through study completion, an average of 90 days
  The Root Mean Squared Error in predicting the greatest diameter stenosis per vessel (Left Main Artery, Left Anterior Descending Artery, Left Circumflex Artery, Right Coronary Artery)

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Mintz, Principal Investigator — CardioVascular Research Foundation
Locations (2):
- United States (2):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Cena Research Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
This data cannot be shared due to individual site data retention policies

REFERENCES:
- [Background] Leasure M, Jain U, Butchy A, Otten J, Covalesky VA, McCormick D, Mintz GS. Deep Learning Algorithm Predicts Angiographic Coronary Artery Disease in Stable Patients Using Only a Standard 12-Lead Electrocardiogram. Can J Cardiol. 2021 Nov;37(11):1715-1724. doi: 10.1016/j.cjca.2021.08.005. Epub 2021 Aug 20. PMID 34419615